CLINICAL TRIAL: NCT01128244
Title: Vitamin B6 Effects on One-Carbon Metabolism
Brief Title: Vitamin B6 Effects for Women Taking Birth Control Pills
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2RO1DKO72398-05
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Vitamin B6 Deficiency
Keywords: oral contraceptives; Vitamin B6; birth control pills; amino acids; Vitamin B6 deficiency; Vitamin B6 deficiency in women on oral contraceptives
MeSH Terms: conditions — Vitamin B 6 Deficiency | interventions — Vitamin B 6; Methionine; Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin B6 Effects in OC Users (Experimental): All subjects will be given an infusion of labeled serine, methionine and leucine prior to vitamin B6 supplementation and after 28 days of treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
  The results from analysis of vitamin B6 and these amino acids in blood will provide us with specific measurements of the rates of two aspects of metabolism (Primary Outcomes 1 and 2) and specific measurements of vitamin B6 nutritional status (Primary Outcomes 3 and 4).
  Interventions: Dietary Supplement: Vitamin B6; Procedure: Infusion of labeled serine, methionine and leucine

INTERVENTIONS:
Dietary Supplement: Vitamin B6 — Subjects will receive vitamin B6 supplementation.
  Other Names: pyridoxine HCl supplement; USP pyridoxine HCL
Procedure: Infusion of labeled serine, methionine and leucine — Subjects will be given an infusion of the stable isotope labeled amino acids, serine, methionine and leucine prior to vitamin B6 supplementation and after 28 days of B6 treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.

SUMMARY:
Chronically inadequate B6 nutritional status is associated with aberrant one-carbon (1C) metabolism and health. Plasma pyridoxal phosphate (PLP) >30 nmol/L often has been considered to be the cutoff indicative of nutritional adequacy, with 20-30 nmol/L considered marginal deficiency; however, the current Recommended Dietary Allowance (RDA) value was based on a more conservative cutoff of 20 nmol/L plasma PLP. As shown by in the investigators preliminary data, biochemical perturbations occur when humans have marginal B6 deficiency consistent with plasma PLP of 20-30 nmol/L. A prospective study also showed that plasma PLP <23.3 nmol/L is associated with 1.8-times higher risk of recurrent venous thromboembolism than those with PLP >23.3 nmol/L. The mechanism by which low B6 intake is associated with risk of vascular disease is not known. Since B6-deficiency has little tendency to raise fasting plasma total homocysteine (tHcy) but yields an elevated tHcy response following a methionine load, low B6 nutriture may lead to repeated transient mild hyperhomocysteinemia following meal consumption. Several reports of associations between elevated plasma C-reactive protein (CRP) and low B6 status have raised the hypothesis that systemic inflammation is prone to occur during B6 deficiency or contributes to low B6 status. The investigators previously found that healthy humans in low B6 status caused by dietary restriction exhibited normal plasma CRP levels. The investigators also postulate that oxidative stress associated with low B6 status, coupled with impaired glutathione synthesis, contributes to such risk. These questions indicate the need for a more thorough understanding of the metabolic changes occurring in low B6 status from marginal B6 intake and from drug interactions such as in women using oral contraceptives.

DETAILED DESCRIPTION:
Potential subjects will undergo a prescreening visit to meet the inclusion criteria, have a history, physical exam and routine labs drawn. The labs will verify the nutritional eligibility of folate, vitamin B12 and vitamin B6. If the inclusion criteria is met then the following will take place.

The subjects will come to the University of Florida (UF) Clinical and Translational Science Institute (CTSI) Clinical Research Center (CRC) for a 9 hour infusion (with stable isotope labeled serine, methionine and leucine) twice during the research study. Once at the start of the study and again at day 29. Blood samples will be taken for metabolite analysis. The infusion of nonradioactive, stable isotope labeled amino acids allows determination of the rate of metabolic reactions in one-carbon metabolism. The results from all subjects' blood analyses will provide us with information about rates of several parts of metabolism and vitamin B6 status.

During the 2-days prior to the infusion a controlled diet will be required. The subjects will be fed at the CTSI CRC. Dietary calculations and formulations will be conducted by using Minnesota Nutrition Data Systems software. Subjects will come to the CRC twice per day where they will meet with staff, consume morning and evening meals, and will be provided a sack lunch and snacks (including weekends). Protein intake will be kept constant.

After the first infusion, all subjects will consume their self-selected usual diets for 28 days along with a commercial B6 supplement providing 10 mg/day. Weekly measurement of blood will be used to verify compliance. All subjects will then consume a 2-day controlled diet at the UF CRC to normalize protein intake, followed by an infusion procedure identical to the first.

During the 4-week supplementation period, all subjects will come to the CRC weekly for weighing, blood samples, and consultation with staff. Careful screening, close monitoring and education of subjects, along with weekly monitoring of blood levels, all contribute to a high degree of compliance.

ELIGIBILITY:
Inclusion Criteria:

* healthy female subjects
* normal screening labs
* normal body weight
* nonpregnant
* Plasma PLP<30nmol/L

Exclusion Criteria:

* history of gastrointestinal surgery
* chronic disease
* vitamin supplementation
* high protein diet
* progesterone
* no smoking
* chronic drug use
* alcoholism
* no vitamin supplementation

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Gregory, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Research Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Gregory JF, DeRatt BN, Rios-Avila L, Ralat M, Stacpoole PW. Vitamin B6 nutritional status and cellular availability of pyridoxal 5'-phosphate govern the function of the transsulfuration pathway's canonical reactions and hydrogen sulfide production via side reactions. Biochimie. 2016 Jul;126:21-6. doi: 10.1016/j.biochi.2015.12.020. Epub 2016 Jan 4. PMID 26765812
- [Derived] Rios-Avila L, Coats B, Ralat M, Chi YY, Midttun O, Ueland PM, Stacpoole PW, Gregory JF 3rd. Pyridoxine supplementation does not alter in vivo kinetics of one-carbon metabolism but modifies patterns of one-carbon and tryptophan metabolites in vitamin B-6-insufficient oral contraceptive users. Am J Clin Nutr. 2015 Sep;102(3):616-25. doi: 10.3945/ajcn.115.113159. Epub 2015 Jul 22. PMID 26201817
- [Derived] Rios-Avila L, Coats B, Chi YY, Midttun O, Ueland PM, Stacpoole PW, Gregory JF 3rd. Metabolite profile analysis reveals association of vitamin B-6 with metabolites related to one-carbon metabolism and tryptophan catabolism but not with biomarkers of inflammation in oral contraceptive users and reveals the effects of oral contraceptives on these processes. J Nutr. 2015 Jan;145(1):87-95. doi: 10.3945/jn.114.201095. Epub 2014 Nov 19. PMID 25527663

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin B6 Effects in OC Users: Subjects will be given an infusion of the amino acids serine, methionine and leucine prior to vitamin B6 supplementation and after 28 days of treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
  Vitamin B6: Subjects will receive vitamin B6 supplementation.
  Infusion of the amino acids, serine, methionine and leucine: Subjects will be given an infusion of the amino acids, serine, methionine and leucine prior to vitamin B6 supplementation and after 28 days of B6 treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
Period: Overall Study
Arm/Group | Vitamin B6 Effects in OC Users
Started | 13
Completed | 10
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Scheduling conflict | 2

BASELINE CHARACTERISTICS:
Groups:
- Vitamin B6 Effects in OC Users: Subjects will be given an infusion of the amino acids, serine, methionine and leucine prior to vitamin B6 supplementation and after 28 days of treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
  Vitamin B6: Subjects will receive vitamin B6 supplementation.
  Infusion of amino acids, serine, methionine and leucine: Subjects will be given an infusion of the amino acids, serine, methionine and leucine prior to vitamin B6 supplementation and after 28 days of B6 treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
Arm/Group | Vitamin B6 Effects in OC Users
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Total Remethylation of Homocysteine
Description: Data from analysis of serine, methionine and leucine in the timed blood samples of all subjects will provide a measurement of the metabolic rate of total remethylation of homocysteine before and after vitamin B6 supplementation.
Time Frame: Blood samples will be taken prior to infusion and at 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7.5, and 9h. Infusions will be conducted at baseline and after 28 days
Population: Women using oral contraceptives exhibiting low vitamin B6 status evaluated at baseline and after vitamin B6 supplementation.
Measure: Mean (Standard Deviation); unit: micromol/(kg x hr)
Groups:
- Total Homocysteine Remethylation Flux: All subjects will be given an infusion of the amino acids serine and methionine prior to vitamin B6 supplementation, and after 28-days of vitamin supplementation. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
Arm/Group | Total Homocysteine Remethylation Flux
Number analyzed (Participants) | 10
micromol/(kg x hr)
  Baseline prior to vitamin supplementation | 6.07 (1.1)
  After 28-days of vitamin supplementation | 5.63 (1.1)
Statistical Analysis 1: Comparison: Total Homocysteine Remethylation Flux; Test type: Superiority or Other; p = 0.20, t-test, 2 sided — Threshold for significance P<0.05; Paired t-test

2. Primary Outcome: Flux of Homocysteine Remethylation From Serine-derived Carbon
Description: Data from analysis of serine, methionine and leucine in the timed blood samples of all subjects will provide a measurement of the metabolic rate of homocysteine remethylation from serine-derived carbon before and after vitamin B6 supplementation. These flux values may be slightly higher than flux of total homocysteine remethylation in Outcome Measure 1 because of the small contribution of methionine salvage to the flux measured in Outcome Measure 2.
Time Frame: as for outcome 1
Population: Women using oral contraceptives and exhibiting low vitamin B6 status.
Measure: Mean (Standard Deviation); unit: micromol/(kg x hr)
Groups:
- Homocysteine Remethylation Flux From Serine: All subjects will be given an infusion of the amino acids serine and methionine prior to vitamin B6 supplementation, and after 28-days of vitamin supplementation. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
Arm/Group | Homocysteine Remethylation Flux From Serine
Number analyzed (Participants) | 10
micromol/(kg x hr)
  Baseline prior to vitamin supplementation | 6.60 (1.9)
  After 28-days of vitamin supplementation | 6.92 (2.2)
Statistical Analysis 1: Comparison: Homocysteine Remethylation Flux From Serine; Test type: Superiority or Other; p = 0.62, t-test, 2 sided — Threshold for significance, P<0.05; Paired t-test

3. Primary Outcome: Fasting Plasma Pyridoxal Phosphate Concentration
Description: For all subjects, the concentration of plasma pyridoxal phosphate in fasting blood samples taken before and after the supplementation period will provide a direct measure of vitamin B6 nutritional status.
Time Frame: Fasting blood samples will be taken at baseline and after 28 days of vitamin B6 supplementation.
Population: Women using oral contraceptives and exhibiting low vitamin B6 status.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Plasma Pyridoxal Phosphate Concentration: Plasma PLP will be measured for all subjects in fasting blood samples obtained at baseline and after 28 days of vitamin B6 supplementation. In addition, all subjects will have weekly weight, blood samples, and visits to the clinic to monitor compliance with the supplementation.
Arm/Group | Plasma Pyridoxal Phosphate Concentration
Number analyzed (Participants) | 10
nmol/L
  Baseline prior to vitamin supplementation | 25.8 (3.6)
  After 28-days of vitamin supplementation | 143 (58)
Statistical Analysis 1: Comparison: Plasma Pyridoxal Phosphate Concentration; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Threshold for significance, P<0.05; Paired t-test

4. Primary Outcome: Fasting Plasma Cystathionine Concentration
Description: For all subjects, the concentration of plasma cystathionine in fasting blood samples taken before and after the supplementation period will provide a functional measure of vitamin B6 nutritional status.
Time Frame: Fasting blood samples will be taken at baseline and after 28 days of vitamin B6 supplementation.
Population: Women using oral contraceptives and exhibiting low vitamin B6 status.
Measure: Mean (Standard Deviation); unit: micromol/L
Groups:
- Plasma Cystathionine Concentration: Plasma cystathionine will be measured for all subjects in fasting blood samples obtained at baseline and after 28 days of vitamin B6 supplementation. In addition, all subjects will have weekly weight, blood samples, and visits to the clinic to monitor compliance with the supplementation.
Arm/Group | Plasma Cystathionine Concentration
Number analyzed (Participants) | 10
micromol/L
  Baseline prior to vitamin supplementation | 0.14 (0.06)
  After 28-days of vitamin supplementation | 0.13 (0.06)
Statistical Analysis 1: Comparison: Plasma Cystathionine Concentration; Test type: Superiority or Other; p = 0.45, t-test, 2 sided — Threshold for significance, P<0.05; Paired t-test

5. Secondary Outcome: Plasma 3-hydroxykynurenine Concentration
Description: For all subjects, analysis of blood samples before and after vitamin B6 supplementation will allow evaluation of discriminating biomarkers using targeted metabolite profile analysis of one-carbon metabolism and tryptophan catabolism constituents. Also, we will conduct exploratory evaluation and potential identification of new biomarkers using metabolomics analysis on subjects before and after vitamin B6 supplementation.
Time Frame: April, 2010 - June, 2014
Population: Women using oral contraceptives and exhibiting low vitamin B6 status.
Measure: Mean (Standard Deviation); unit: microl/L
Groups:
- Secondary Analysis: Plasma 3-hydroxykynurenine Concentration: Plasma 3-hydroxykynurenine concentration will be measured for all subjects in fasting blood samples obtained at baseline and after 28 days of vitamin B6 supplementation. In addition, all subjects will have weekly weight, blood samples, and visits to the clinic to monitor compliance with the supplementation.
Arm/Group | Secondary Analysis: Plasma 3-hydroxykynurenine Concentration
Number analyzed (Participants) | 10
microl/L
  Baseline prior to vitamin supplementation | 25.9 (14.0)
  After 28-days of vitamin supplementation | 27.3 (14.0)
Statistical Analysis 1: Comparison: Secondary Analysis: Plasma 3-hydroxykynurenine Concentration; Data were analyzed by paired t-test adjusted for multiple testing by Sidak methods; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Data were analyzed by paired t-test adjusted for multiple testing by Sidak methods; Test of treatment effect. = 0.05

ADVERSE EVENTS:
Groups:
- Vitamin B6 Effects in OC Users: Subjects will be given an infusion of the amino acids serine and methionine prior to vitamin B6 supplementation and after 28 days of treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
  Vitamin B6: Subjects will receive vitamin B6 supplementation.
  Infusion of amino acids, serine, and methionine: Subjects will be given an infusion of the amino acids, serine, and methionine prior to vitamin B6 supplementation and after 28 days of B6 treatment. In addition, they will receive a special diet 2 days prior to the infusion and will have weekly weight, blood, and visits to the clinic.
Arm/Group | Vitamin B6 Effects in OC Users
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin B6 Effects in OC Users (N=13)
Vasovagal reaction (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Secondary Outcome Measure(s): 5. Data Not Reported Exploratory Metabolite Profile and Metabolomics Analysis. The Analysis from the lab was delayed due to circumstance beyond our control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No